CLINICAL TRIAL: NCT03410277
Title: Measurement of Glucose Homeostasis in Human Brain by NMR: Effect of Recurrent Hypoglycemia on Type 1 Diabetes (Aim 1)
Brief Title: Recurrent Hypoglycemia in Type 1 Diabetes (Aim 1)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: MED-2017-26317
Record Dates: First submitted 2018-01-18; First posted 2018-01-25 (Actual); Last update posted 2024-05-03 (Actual); Status verified 2024-05

CONDITIONS: Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- All Subjects (Experimental): Experimental hypoglycemia
  Interventions: Other: Experimental hypoglycemia

INTERVENTIONS:
Other: Experimental hypoglycemia — Experimental hypoglycemia with and without MRI

SUMMARY:
This study will explore the cerebral mechanisms of impaired awareness of hypoglycemia (IAH) in type 1 diabetics following exposure to experimental recurrent hypoglycemia (HG). To induce IAH, patients with T1D identified to have normal awareness of hypoglycemia (NAH) will undergo three 2-hour long hypoglycemic clamps. Neurochemical profiles will be measured by high field MRS before and after induction of IAH. Subject glycemic variability for 2 weeks and activity/sleep for 1 week before each study will be monitored as all factors have been shown to alter responses to HG.

DETAILED DESCRIPTION:
The long-term goal of this project is to identify how recurrent hypoglycemia (HG) leads to the clinical syndrome of impaired awareness of hypoglycemia (IAH) in type 1 diabetes (T1D). This study will test the hypothesis that recurrent HG in T1D leads to an upregulation in brain glucose transport and alterations in glutamatergic and GABAergic tone. The investigators will use MRS methodology that permits evaluation of cerebral cortex and hypothalamus in the same session to simultaneously evaluate the cerebral correlates/mediators of impaired awareness and impaired counterregulatory hormone responses (CRR). High MR data quality and reproducibility will be ensured by using high field MR scanners and technical advances (automated voxel placement, real-time voxel position, frequency, shim updates). Continuous glucose monitoring and actigraphy will be used to chronicle glucose variability and activity/exercise/sleep in the weeks before each experiment to assess the impact of these variables on IAH.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes diagnosed on clinical or laboratory grounds
* Diabetes duration 2 - 30 years
* Hemoglobin A1C <8.5%

Exclusion Criteria:

* Impaired awareness of hypoglycemia as determined by the Cox and Gold questionnaires
* Pregnant or plan to become pregnant during the study period
* Uncontrolled hypertension (blood pressure > 145/95 mmHg at screening)
* Evidence of autonomic neuropathy (presence of orthostatic hypotension or history of gastroparesis)
* Proliferative retinopathy
* Impaired kidney function (GFR < 45)
* History of myocardial infarction, stroke, seizures, neurosurgical procedures, major depression requiring hospitalization within the last 5 years, arrhythmias
* Current substance abuse
* Use of drugs that can alter glucose metabolism including but not limited to glucocorticoids and niacin, and excluding insulin and glucose lowering drugs used to treat diabetes, as determined by a clinician
* Inability to undergo MRI scanning, including but not limited to unable to remain still in an MRI scanner for more than 30 minutes, claustrophobia, presence of paramagnetic substances or pacemakers in body, weight over 300 lbs

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2018-05-24 (Actual); Primary Completion 2024-03-31 (Actual); Study Completion 2024-03-31 (Actual)

PRIMARY OUTCOMES:
Neurochemical response to HG before and after induction of IAH | 240 Minutes
  The difference in neurochemical response (GABA, glutamate, and glucose) to HG during the first clamp study compared to the neurochemical response to HG after the induction of IAH as determined by the last clamp.

SECONDARY OUTCOMES:
Antecedent glycemia concentration | 16 days
  The difference in antecedent glycemia concentration associated with the differences seen in the primary outcome.
Antecedent physical activity | 16 days
  The difference in antecedent physical activity associated with the differences seen in the primary outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth R Seaquist, MD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No